CLINICAL TRIAL: NCT04183153
Title: Endo-Connectome Study
Brief Title: Neuroendocrine Mapping of the Cerebral Cortex
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left lab
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 53928
Record Dates: First submitted 2019-11-25; First posted 2019-12-03 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Arm (Experimental)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Participants will receive repetitive transcranial magnetic stimulation (rTMS) to determine if stimulating areas with activating functional connectivity will activate the hypothalamus and in turn, have a measurable effect on hormone levels.

SUMMARY:
This study is investigating brain regions that share functional connectivity with the hypothalamus and the stimulation of those regions using repetitive transcranial magnetic stimulation (rTMS) to activate the hypothalamus indirectly. The goal of this study is to determine the effectiveness of rTMS in influencing the hypothalamus to better understand the mechanisms between it and the neuroendocrine processes it controls.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-55
* Gender: Females and Males
* Weight: Less than 280 pounds
* Mobile
* Normal vision with corrective lenses if necessary
* Fluent in English (written and spoken)

Exclusion Criteria:

* History of epilepsy/seizures (including history of withdrawal/provoked seizures)
* Metal implant in brains (e.g. deep stimulation), cardiac pacemaker, or cochlear implants
* Shrapnel or any ferromagnetic item in the head
* Showing symptoms of withdrawal from alcohol or benzodiazepines
* Current severe insomnia (must sleep a minimum of 4 hours the night before stimulation)
* Migraine or significant headaches
* Shoulder or neck stiffness
* Over 280 pounds
* In-dwelling ferrous metals
* Left handed
* Abnormal hearing
* Abnormal vision that cannot be corrected with lenses
* Claustrophobia
* Illicit drug use
* Psychotropic medication use
* Marijuana and/or nicotine use
* Psychiatric or neurological conditions
* Endocrine conditions
* History of head trauma with loss of consciousness

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma GnRH levels resulting from hypothalamus activation via LC-MS | 3 hours
  Measure levels of the gonadotropin-releasing hormone (GnRH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma vasopressin levels via LC-MS | 3 hours
  Measure levels of the vasopressin hormone in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma oxytocin levels via LC-MS | 3 hours
  Measure levels of the oxytocin hormone in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma TRH levels via LC-MS | 3 hours
  Measure levels of the thyrotropin-releasing hormone (TRH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma CRH levels via LC-MS | 3 hours
  Measure levels of the corticotropin-releasing hormone (CRH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma somatostatin levels via LC-MS | 3 hours
  Measure levels of the somatostatin hormone, or growth hormone-inhibiting hormone (GHIH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma PRLH levels via LC-MS | 3 hours
  Measure levels of the prolactin-releasing hormone (PRLH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma FSH levels via LC-MS | 3 hours
  Measure levels of the follicle-stimulating hormone (FSH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma LH levels via LC-MS | 3 hours
  Measure levels of the luteinizing hormone (LH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma ACTH levels via LC-MS | 3 hours
  Measure levels of the adrenocorticotropic hormone (ACTH) in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation
Plasma cortisol levels via LC-MS | 3 hours
  Measure levels of the cortisol hormone in blood plasma through liquid chromatography-mass spectrometry (LC-MS) resulting from hypothalamus and neuroendocrine activation

SECONDARY OUTCOMES:
Blood pressure via sphygmomanometer | 3 hours
  Measure systolic and diastolic blood pressure (BP) with a sphygmomanometer as a secondary measure of hypothalamic response
Heart rate via pulse oximeter | 3 hours
  Measure heart rate (HR) with a pulse oximeter as a secondary measure of hypothalamic response

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sudheimer, Ph.D., Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No